CLINICAL TRIAL: NCT01876628
Title: A Double Blind Randomised Control Trial to Measure the Effect of the Addition of Clindamycin to Flucloxacillin for the Treatment of Limb Cellulitis
Brief Title: Adjunctive Clindamycin for Cellulitis: C4C Trial.
Acronym: C4C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: University of Bristol (Other); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4C-4078; 2013-001218-14 (EudraCT Number)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Cellulitis
Keywords: Clindamycin; Cellulitis; Flucloxacillin; Group A streptococcus; Staphylococcus aureus
MeSH Terms: conditions — Cellulitis; Staphylococcal Infections | interventions — Floxacillin; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flucloxacillin and Placebo oral capsule (Placebo Comparator): Intravenous or oral Flucloxacillin with a Placebo oral capsule
  Interventions: Drug: Flucloxacillin; Drug: Placebo oral capsule
- Flucloxacillin and Clindamycin (Active Comparator): Intravenous or oral Flucloxacillin with Clindamycin oral capsule
  Interventions: Drug: Flucloxacillin; Drug: Clindamycin

INTERVENTIONS:
Drug: Flucloxacillin — Intravenous or oral Flucloxacillin. Minimum dose 500mg four times each day. Target duration 5 days less pre-recruitment beta-lactam duration.
  Other Names: Floxapen; Fluclomix; Ladropen
Drug: Clindamycin — Clindamycin dose 300mg four times each day for 2 days, within 48 hours of commencing flucloxacillin. Clindamycin is over-encapsulated and externally identical to placebo.
  Other Names: Dalacin C; Daclin; Cleocin
  Arms: Flucloxacillin and Clindamycin
Drug: Placebo oral capsule — Placebo is externally identical to the over-encapsulated clindamycin and is taken four times each day for 2 days
  Arms: Flucloxacillin and Placebo oral capsule

SUMMARY:
The aim of this study is to see whether the addition of Clindamycin, a protein inhibiting antibiotic, to the standard antibiotic treatment of limb cellulitis, with Flucloxacillin, results in less tissue damage and a more rapid resolution of both systemic and local features, in a cost-effective manner. This study is a randomised controlled trial comparing Clindamycin with placebo.

DETAILED DESCRIPTION:
Criteria to be used to assess tissue damage and clinical response:

1. Fever, tachycardia, neutrophil count, urea and other laboratory parameters at five and ten days post first dose of clindamycin
2. Limb swelling (by the measurement of limb circumference), skin surface temperature and tissue damage (by the proportion of the limb affected)
3. Document the duration between initial systemic features and the development of local signs
4. Examine the effect of the duration between systemic and local features and first dose of flucloxacillin on the subsequent duration and severity of cellulitis
5. Examine the effect of duration between the first dose of flucloxacillin and the first dose of clindamycin on the subsequent duration and severity of cellulitis
6. Identify and quantify possible side effects of clindamycin

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 or over who have a diagnosis of cellulitis of a single, upper or lower, limb
* Who are able to understand the study and give consent
* Who are able to take oral medication

Exclusion Criteria:

* Patients with a confirmed history of penicillin, flucloxacillin or clindamycin allergy
* Patients known to be colonised with Methicillin-resistant Staphylococcus aureus or Methicillin-resistant Staphylococcus aureus isolated from wound within the last year
* Patients unable to take oral medication
* Previous history of Clostridium difficile colitis
* Clindamycin taken within the last 30 days
* Clinically unstable
* Unable to understand the study or give consent
* Any doubt over the certainty of the diagnosis of cellulitis
* Patients taking any drug that is incompatible with either flucloxacillin or clindamycin
* Pre-existing diarrhoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Improvement based on a composite of systemic and local features | Day 5
  Temperature less than 37.5 degrees centigrade, reduction in limb swelling and reduction in skin temperature

SECONDARY OUTCOMES:
Decrease in pain | Day 10
  Assessed using a visual analogue score
Quality of life | Day 30
  Assessment based on a questionnaire plus return to work or normal activities and absence of increased side-effects.
Physiological recovery | Day 10
  Resolution of systemic features, composite inflammatory markers and recovery of renal function.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Bristol NHS Foundation Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Brindle R, Williams OM, Davies P, Harris T, Jarman H, Hay AD, Featherstone P. Adjunctive clindamycin for cellulitis: a clinical trial comparing flucloxacillin with or without clindamycin for the treatment of limb cellulitis. BMJ Open. 2017 Mar 17;7(3):e013260. doi: 10.1136/bmjopen-2016-013260. PMID 28314743